CLINICAL TRIAL: NCT06923787
Title: Effect of Perioperative Intravenous Infusion of Lidocaine on the Postoperative Course and the Immune Response in Patients Undergoing Surgery for Colon Cancer - the PILDI Study
Acronym: PILDI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ORI2025-016; 2025-521808-22-01 (EU CTIS Number)
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Double-blind randomized trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidokaine arm (Active Comparator): Patients who will receive intravenous lidocaine.
  Interventions: Drug: Lidocaine
- Placebo arm (Placebo Comparator): Patients who will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — intravenous infusion of lidocaine
  Arms: Lidokaine arm
Drug: Placebo — saline solution intravenous infusion
  Arms: Placebo arm

SUMMARY:
There are very few data in the literature on changes in inflammatory markers when lidocaine is administered perioperatively in patients with colorectal cancer. In patients undergoing surgery for colon cancer, the aim is to conduct a double-blind placebo-controlled study to determine differences in levels of pro-inflammatory markers, postoperative pain and opioid analgesic consumption in the first two days after surgery, and the time to first postoperative bowel movement. Groups of patients receiving perioperative lidocaine infusion, high dose dexamethasone or placebo will be compared.

DETAILED DESCRIPTION:
In 80% of cancer patients, surgery is indicated during treatment. The choice of anasthetic technique can indirectly influence the patient's inflammatory and immune systems. Although a large body of data on the association between surgical stress and anasthesia in in vitro tumor models is already available, the importance of the individual drugs used during anasthesia on the inflammatory response and the post-operative course of patients is not yet fully understood, and further research is needed in this area.

There is increasing evidence that perioperative intravenous infusion of lidocaine has analgesic, prokinetic and anti-inflammatory properties in patients treated with surgical procedures. A significant number of studies have confirmed the positive effects of intravenous lidocaine infusion on reducing postoperative pain and reducing perioperative opioid consumption. In recent years, a growing number of studies have investigated the positive effects of lidocaine infusion on promoting peristalsis and faster recovery after surgery and on reducing the perioperative inflammatory response. This effect is also beneficial after colon surgery.

Inflammation is particularly detrimental in cancer patients as it may be associated with more frequent postoperative complications, slower recovery, and poorer cancer outcome (recurrence and/or survival), irrespective of the incidence of perioperative complications.

Surgical stress may promote tumor sequelae in several ways: ischemia and reperfusion injury, sympathetic nervous system activation, inflammation, systemic hypercoagulable state, immune suppression and the effects of anesthetics.

Proinflammatory markers, postoperative pain, opioid consumption, time to first postoperative bowel movement, and the effect on postoperative course in groups of patients receiving perioperative infusion of lidocaine or placebo have not yet been investigated in a double-blind placebo-controlled study. The data generated in this study may represent an important scientific contribution with a positive impact on the management of patients undergoing surgery for colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* colon cancer of any stage of the disease for which elective laparoscopic colon resection and colonic anastomosis will be performed,
* age of patients between 18 and 80 years,
* low to moderate risk of anesthesia (ASA up to and including 3),
* ability to understand the study and to sign an informed consent to participate in the study

Exclusion Criteria:

* patients receiving neoadjuvant chemotherapy,
* pregnancy or breastfeeding,
* known allergy to lidocaine
* cardiac rhythm disturbances (bradycardia < 45 beats/min, complete heart block, use of group III antiarrhythmics),
* status post cardiac arrest,
* porphyria,
* myasthenia gravis,
* severe hepatic impairment (cirrhosis, ascites, bleeding disorders, jaundice, encephalopathy),
* renal disease (hamodialysis, creatinine clearance <30 mL/min),
* epilepsy,
* active infection,
* presence of viral or systemic fungal disease,
* uncontrolled psychotic state,
* ulcerative gastric or duodenal disease,
* chronic corticosteroid therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-03 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Difference in opioid use in 24 hours after surgery between arms | 24 hours after surgery
  Patients who receive a perioperative infusion of lidocaine will have lower need for opioid consumption oppose to placebo arm

SECONDARY OUTCOMES:
Time to bowel movement after surgery | observation within 30 days after surgery
  Patients receiving a perioperative infusion of lidocaine will have a shorter time to first postoperative bowel movement than patients receiving placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Nikola Bešić, MD, Principal Investigator — Institute of Oncology Ljubljana
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No